CLINICAL TRIAL: NCT06345677
Title: An Exploratory, Prospective, Multicenter, Randomized, Double Blind, Placebo + Sham Device Controlled, Study to Assess the Safety, Usability, and Initial Efficacy of the ViXe Combination for Intravesical Administration of XEOMIN® in the Treatment of Female Patients With Idiopathic Overactive Bladder (OAB)
Brief Title: Clinical Trial for the Assessment of Safety, Usability and Efficacy of the Vixe Combination for OAB in Female Subjects
Acronym: XAVIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vensica Therapeutics Ltd. (Industry)
Collaborators: Blueclinical, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ViXe-CLP-0002
Record Dates: First submitted 2024-02-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ViXe Combination (Experimental): This arm includes a combination of the Xeomin medication, a generic of the Botulinium Toxin A drug that is not currently approved for this indication, and the Vibe medical device, an experimental device for the delivery of Botulinium Toxin to the bladder for overactive bladder
  Interventions: Combination Product: ViXe Xombination
- Placebo + Sham (Placebo Comparator): The placebo that will be used in the study is identical in its physical properties to the investigational drug and will be used in the same manner as the active drug. Sham procedure will include all the steps for device preparation and activation, without the actual transmission of ultrasound eneregy to the participant.
  Interventions: Combination Product: Placebo + Sham

INTERVENTIONS:
Combination Product: ViXe Xombination — Combination of Xeomin and the ultrasound based delivery system (Vibe) for intravesical administration of the drug in a minimally invasive procedure
  Arms: ViXe Combination
Combination Product: Placebo + Sham — Placebo identical in package and appearance to Xeomin together with all steps of Vibe device preparation and activation, but without the actual operation of the ultrasound energy
  Arms: Placebo + Sham

SUMMARY:
The goal of this interventional clinical trial is to assess the safety, usability and initial efficacy of Xeomin and Vibe combination (ViXe) compared to placebo + sham in female subjects with idiopathic Overactive Bladder. The main question[s] it aims to answer are: • The rate of device and drug related serious adverse events during treatment and throughout the follow up period • Investigator, subject and technician satisfaction from treatment, and • Assess the initial efficacy of the drug-device combination compared to placebo-sham combination. Participants will be treated a single time with the ViXe combination and will be followed up for a period of 12 weeks, during which they will visit the clinic after 2, 6 and 12 weeks. Participants will complete a 3-day voiding diary prior to the 6- and 12-week FU visit.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18 and 80 years at the time of signing the informed consent.
* Signed written informed consent.
* Diagnosis of OAB for at least 6 months prior to screening, determined by documented subject history.
* At least 8 voiding episodes/day based on 3-consecutive days voiding diary at screening.
* OAB with at least 6 leaking episodes associated with urgency (UUI), and at least one episode per day demonstrated on 3-consecutive days voiding diary.
* Subject is mentally competent with the ability to understand and comply with the requirements of the study.
* Subject is willing and able to initiate self-catheterization post treatment, if required.
* Subject with inadequate response to conservative medication treatment/s as defined by the investigator.
* Subject agrees to attend all follow-up evaluations and is willing and capable to fill out voiding diaries and questionnaires completely and accurately and is willing to complete required exams and tests.
* Females with childbearing potential must have a negative pregnancy test and must practice an acceptable method of birth control, from at least 4 weeks before treatment until 12 weeks after treatment

Exclusion Criteria:

* Previous participation in another study with any investigational drug or device within the past 90 days.
* Allergy to Botulinum neurotoxin type A or any of the other ingredients and components of this device or the drug
* Subject with OAB caused by neurological conditions (i.e., Myasthenia Gravis, ALS, Eaton-Lambert Syndrome, etc.)
* Any neurological disease or disorder including Alzheimer's, Parkinson, MS, stroke (CVA), neuropathy or injury resulting in neuropathy.
* Subject currently under treatment with biofeedback, pelvic muscle rehabilitation, pelvic floor physical therapy. If willing to discontinue will be allowed to participate after 4 weeks of wash out. Self-Kegels exercises are allowed.
* Bleeding disorders or treatment with anticoagulants, antiplatelet (except acetylsalicylic acid), or thrombolytic medications within 14 days prior to screening.
* Subjects with compromised respiratory function or dysphagia.
* Current or planned treatment with drugs that interfere with neuromuscular transmission (e.g., aminoglycoside, polypeptide antibiotics, lincomycin antibiotics, or aminoquinolines)
* Subject with known polyuria/polydipsia with 24-hour total volume void > 3000 ml.
* Subject with PVR ≥ 200 ml based on bladder ultrasound at screening visit.
* Current or recurrent urinary tract infection (3 or more infections in the last 6 months), or presence of urinary fistula per physical examination, or known significant urinary tract obstruction or urethral stricture.
* Subject who received botulinum toxin injections within the past 8 months.
* Subject with predominant stress incontinence based on MESA incontinence score and/or voiding diary at screening.
* BMI ≥ 35 kg/m2.
* If used, should be on stable doses of diuretics for the past 3 months.
* Subjects who have any implanted electronic devices (a pacemaker, for example), permanent or transient, that cannot be removed prior to the treatment.
* Subjects who have received tibial or sacral nerve stimulation (SNS) any time in the past or percutaneous tibial nerve (PTNS) in the last 3 months.
* Previous urinary incontinence surgery or prolapse surgery or de novo urinary incontinence post-surgery within the last 12 months.
* Any spinal surgery within the last 12 months.
* Previous abdominoperineal resection of the rectum or previous radical hysterectomy.
* Diagnosis of interstitial cystitis or bladder pain syndrome as defined by either American Urological Association (AUA) or European Association of Urology (EAU) guidelines.
* History of evidence of anatomic pelvic, urological or urogenital abnormality according to investigator's discretion.
* If used, subjects should be on stable dose of antimuscarinics and/or beta-3 adrenergic agonists for at least 3 months prior to enrolment and agree to remain on stable medication consumption until the 12-weeks follow-up visit.
* If used, subjects should be on a stable dose of tricyclic antidepressants, Selective Serotonin Reuptake Inhibitors (SSRI) and Serotonin-Norepinephrine Reuptake Inhibitors (SNRI) for at least 3 months prior to enrolment and agree to remain on stable medication consumption until the 12 weeks follow-up visit.
* Subject with abnormal renal function defined by estimated glomerular filtration rate (eGFR) of 30 ml/min or less.
* History of pelvic radiotherapy or chemotherapy for pelvic malignancies.
* Diabetes with peripheral nerve neuropathy or severe uncontrolled diabetes (with HbA1C > 7.5%).
* Uterine prolapse, cystocele, enterocele or rectocele past the hymen.
* Deemed unsuitable for enrollment by the investigator based on history or physical examination.
* Any psychiatric or personality disorder at the discretion of the study physician.
* Any severe or uncontrolled systemic disease (e.g., cardiac, renal, pulmonary, hepatic, or gastrointestinal), malignant tumor, or medical history of HIV infection, or any findings from laboratory or physical examination performed at screening at the discretion of the investigator
* Subject is breastfeeding
* Drug or alcohol abuse

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events Rate | 12 weeks
  Incidence of drug and device related adverse events from treatment to 12-weeks post treatment
Usability and ease-of-use perception by investigator, subject and technician | Procedure
  Satisfaction of investigator, participant and technicain from the treatment, as assessed by the sponsor designed usability questionnaire.
  Investigator's questionnaire consists of 43 questions on a scale of 1-7 each (total range 43-301). The higher the total score, the better the investigator satisfaction. Subject usability questionnaire consists of 11 questions on a scale of 0-10 (total range 0-110). Thr higher the score, the more statisfied the subject from the treatment. Technician's questionnaire consists of yes/no questions only.

SECONDARY OUTCOMES:
Daily Urgency Urinary Incontinence | 12 weeks
  Mean change from baseline in the average number of daily Urgency Urinary Incontinence (UUI) Episodes at 6 and 12-weeks post treatment based on a 3-day voiding diary
Total Daily Episodes | 12 weeks
  Mean change from Baseline in the average number of daily voiding episodes at 6 and 12-weeks post treatment based on a 3-day voiding diary
Urinary Urgency | 12 weeks
  Mean Change from baseline in Urinary grade 3 or 4 Urgency Episodes at 6 and 12-weeks post treatment based on a 3-day voiding diary
Voiding Leaks | 12 weeks
  Mean change from baseline in Number of large leaks at 6 and 12-weeks post treatment based on a 3-day voiding diary
Quality of Life Queationnsaire | 12 weeks
  Change from baseline in OAB-q (Overactive Bladder - quality) total score at week 12. OAB-q is a two-domain questionnaire (symptom bother and health related quality of life), each of which is a 100-point scale. Higher scores reflect higher quality of life.
Nocturia | 12 weeks
  Mean change from baseline in the average number of daily Nocturia episodes at 6 and 12-weeks post treatment based on a 3-day voiding diary

CONTACTS AND LOCATIONS:
Overall Officials: Palma dos Reis, Dr, Principal Investigator — Principal investigator at CHLN
Locations (8):
- Portugal (8):
  - CHUC, Coimbra
  - HSOG, Guimarães
  - CHLN, Lisbon
  - CHUSJ, Porto
  - Hospital Lusíadas, Porto
  - Hospital Prelada, Porto
  - Hospital Luz Setúbal, Setúbal
  - CHVNG, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: No
All subjects will be assigned a unique study code that will not enable anyone outside of the study team on site to identify them. No personal data will be colected during the study other than date of birth.